CLINICAL TRIAL: NCT00203684
Title: The Effects of Different Sized Inhaled Corticosteroids on Peripheral Lung Inflammation in Asthma Assessed Through Lung Tissue Samples (SMART Protocol)
Brief Title: Mentored Patient-Oriented Research Career Development Award
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5K23RR018538-03 (NIH); NIH grant #5K23RR018538-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2017-02

CONDITIONS: Asthma; Distal Lung Inflammation
MeSH Terms: conditions — Asthma | interventions — flunisolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Small particle corticosteroid (Other): In the first phase, the investigators will collect baseline information about subjects while they are using placebo (inactive substance). In the second phase, subjects will take the small particle corticosteroid that should reach both the large and small airways (Flunisolide-HFA).
  Interventions: Drug: Flunisolide-HFA
- Large particle corticosteroid (Other): In the first phase, the investigators will collect baseline information about subjects while they are using placebo (inactive substance). In the second phase, subjects will take the large particle corticosteroid that should only reach the large airways (Flunisolide-CFC).
  Interventions: Drug: Flunisolide-CFC

INTERVENTIONS:
Drug: Flunisolide-HFA — an inhaled, small particle corticosteroid that should reach both the large and small airways (Flunisolide-HFA)
  Other Names: Small particle corticosteroid
  Arms: Small particle corticosteroid
Drug: Flunisolide-CFC — an inhaled corticosteroid that has a large particle size and should only reach the large airways (Flunisolide-CFC)
  Other Names: Large particle corticosteroid
  Arms: Large particle corticosteroid

SUMMARY:
Asthmatics have inflammation in the large airways (tubes through which air travels in and out of the lungs). The large airways are located in the central lung. New research shows that asthmatics also have inflammation in the small airways. The small airways are located in the peripheral lung (the parts of the lung away from the central lung).

Until now, most of the inhaled medications available have been made up of big particles that never reach the peripheral lung. The purpose of this study is to try to measure the level of inflammation in the peripheral lung in asthmatics and see if this inflammation can be decreased with different types of inhaled corticosteroids. The investigators will check airway inflammation before and after use of an inhaled corticosteroid that has a large particle size and should only reach the large airways (Flunisolide-CFC), and before and after use of an inhaled, small particle corticosteroid that should reach both the large and small airways (Flunisolide-HFA).

Subjects will make 6 study visits over two phases of the study. In the first phase, the investigators will collect baseline information about subjects while they are using placebo (inactive substance). In the second phase, subjects will take either the large or small particle corticosteroid.

Visits will involve questionnaires and various tests measuring lung function (such as spirometry, forced oscillation, and methacholine challenge). Exhaled nitric oxide will be measured as an indication of inflammation. Subjects will also measure and make note of lung function at home twice daily using a peak expiratory flow meter. Two of the visits will involve fiberoptic bronchoscopy so that the investigators may collect cells and tissue samples without surgery. Another two of the visits will involve the use of high resolution computed tomography (HRCT) scans to indirectly evaluate disease in distant parts of the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years. Younger subjects are excluded due to greater concerns with respect to risks from radiation and bronchoscopy in children; older subjects due to greater risks of bronchoscopy.
* Mild to moderate persistent asthma (forced expiratory volume in 1 second [FEV1] greater than or equal to 70% predicted {Hankinson, 1999 #266}; PC20 less than or equal to 8 mg/ml) and currently using only short acting inhaled beta agonists as needed for control of asthma symptoms.

Exclusion Criteria:

* The use of the following medications will exclude subjects from entering the study:

  * Oral or parenteral steroids within 6 months
  * Inhaled corticosteroids within 3 months
  * Antileukotrienes, b-adrenergic blocking agents, inhaled cromolyn sodium or nedocromil, macrolide antibiotics, or investigational drugs within 1 month
  * Drugs or exposures which, in the opinion of the investigators, could influence study results
* Tobacco within 1 year or less than or equal to 5 pack years.
* Pregnant women, lactating women, or women of childbearing age not willing to take precautions to avoid becoming pregnant during the study.
* Subjects with upper respiratory infection or receiving an influenza vaccine within 6 weeks of the study.
* Subjects with a history of allergy or adverse reaction to inhaled beta agonists or methacholine.
* Subjects with clinically significant evidence of cardiovascular, central nervous system, endocrine, gastrointestinal, hematopoietic, hepatic, psychiatric, or respiratory (other than asthma) disease

Eligibility will be determined by an investigator using the above inclusion/exclusion criteria.

No subjects will be excluded based on race or gender. Subjects must be between 18 and 50 in order to avoid greater risks of bronchoscopy and, in those under 18, exposure to radiation. To avoid risks, women will not be enrolled if pregnant, lactating or of childbearing potential and unwilling to undertake appropriate precautions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Zeidler, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Asthma and Cough Center, Los Angeles, California, United States